CLINICAL TRIAL: NCT05664750
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Active-Controlled Phase III Study to Compare the Efficacy and Safety of Passive Immunization With TNM002 Injection and Human Tetanus Immunoglobulin as Prophylaxis Against Tetanus
Brief Title: Study to Compare the Efficacy and Safety of Passive Immunization With TNM002 Injection and Human Tetanus Immunoglobulin as Prophylaxis Against Tetanus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNM002-301
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-10

CONDITIONS: Tetanus
Keywords: Tetanus; Prophylaxis
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Intervention Model Description: Participants will be randomized and receive a single intramuscular injection (IM) gluteal injection of TNM002 or human tetanus immunoglobulin (HTIG).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNM002 (Experimental): If randomized to TNM002, participant will receive a single IM gluteal injection of TNM002
  Interventions: Drug: TNM002
- Human tetanus immunoglobulin (HTIG) (Active Comparator): If randomized to HTIG, participant will receive a single IM gluteal injection of HTIG
  Interventions: Drug: Human tetanus immunoglobulin (HTIG)

INTERVENTIONS:
Drug: TNM002 — Dosage Form: Injection, solution
  Route of administration: IM gluteal injection
  Arms: TNM002
Drug: Human tetanus immunoglobulin (HTIG) — Dosage Form: Injection, solution
  Route of administration: IM gluteal injection
  Arms: Human tetanus immunoglobulin (HTIG)

SUMMARY:
TNM002 Injection is a recombinant fully human native monoclonal antibody (mAb) against tetanus toxin and is currently under development for indication of prophylaxis against tetanus.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female adults aged ≥ 18 years;
2. Participants with dirty or contaminated wounds caused by various injury who require passive immunization as prophylaxis against tetanus;
3. Participants who provide signed written informed consent form.

Exclusion Criteria:

1. Known or suspected allergy to the investigational product or its excipients, or have a history of allergy to human immunoglobulin products or other therapeutic monoclonal immunoglobulins;
2. Suspect or diagnosed as tetanus;
3. Previously diagnosed as Immunoglobulin A (IgA) deficiency with anti-IgA antibodies
4. Prior vaccination history of ≥ 3 doses of tetanus toxoid or tetanus toxoid- containing vaccine;
5. Current alcohol abuse, drug abuse or drug addiction

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with an increase of anti-tetanus neutralizing antibody titers (∆ titers) over protective level. | Baseline up to 12 hours after receipt of study drug

SECONDARY OUTCOMES:
Tetanus protection rate (1 - tetanus incidence) | Up to 28 days after receipt of study drug

OTHER OUTCOMES:
Incidence of adverse events (AEs) | Up to 105 days after receipt of study drug
Incidence of treatment related adverse events (AEs) | Up to 105 days after receipt of study drug
Incidence of serious adverse events (SAEs) | Up to 105 days after receipt of study drug
The number and percentage of subjects with abnormal hematology tests | Up to 90 days after receipt of study drug
  The hemotology tests include red blood cell count, hemoglobin, platelet count, white blood cell count, absolute neutrophil count, neutrophil percentage, absolute lymphocyte count, lymphocytes percentage, absolute monocyte count, and hematocrit
The number and percentage of subjects with abnormal serum chemistry tests | Up to 90 days after receipt of study drug
  The serum chemistry tests include total protein, albumin, sodium, potassium, chloride, calcium, glucose, aspartate aminotransferase, alanine aminotransferase, total bilirubin, direct bilirubin, urea (blood urea nitrogen) and creatinine
The number and percentage of subjects with abnormal urinalysis tests | Up to 90 days after receipt of study drug
  The urinalysis tests include protein, glucose, urobilinogen, urine occult blood, red blood cell and white blood cell
The number and percentage of subjects with abnormal vital signs | Up to 90 days after receipt of study drug
  The vital signs include blood pressure, pulse rate, respiratory rate, and body temperature
The number and percentage of subjects with abnormal physical examination | Up to 90 days after receipt of study drug
  The physical examination includes skin, lymph nodes, eyes, head and neck, chest, abdomen, spine, extremities.
The number and percentage of subjects with abnormal 12-lead electrocardiogram (ECG) | Up to 90 days after receipt of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Chuanlin Wang, MD, Principal Investigator — Peking University People's Hospital; Shengyi Wang, Study Director — Zhuhai Trinomab Pharmaceutical Co., Ltd.
Locations (28):
- China (28):
  - Hefei First People's Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Liuzhou Worker's Hospital - Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi
  - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Zhejiang Provincial People's Hospital, Hangzhou, Hangzhou
  - The Central Hospital of Wuhan, Tongji Medical College Huazhong University of Science&Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Affiliated Nanhua Hospital, University of South China, Hengyang, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - PKUCare Luzhong Hospital, Zibo, Shandong
  - The First People's Hospital of Jinzhong, Jinzhong, Shanxi
  - Shanxi Academy of Medical Sciences - Shanxi Bethune Hospital (Shanxi Dayi Hospital), Taiyuan, Shanxi
  - Yuncheng Central Hospital - East Campus, Yuncheng, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang CL, Liu S, Shao ZJ, Yin ZD, Chen QJ, Ma X, Ma C, Wang Q, Wang LH, Deng JK, Li YX, Zhao ZX, Wu D, Wu J, Zhang L, Yao KH, Gao Y, Xie X. [Guidelines for the use of post-traumatic tetanus vaccines and passive immune preparation]. Zhonghua Yu Fang Yi Xue Za Zhi. 2019 Dec 6;53(12):1212-1217. doi: 10.3760/cma.j.issn.0253-9624.2019.12.005. Chinese. PMID 31795577
- [Background] Roper MH, Vandelaer JH, Gasse FL. Maternal and neonatal tetanus. Lancet. 2007 Dec 8;370(9603):1947-59. doi: 10.1016/S0140-6736(07)61261-6. PMID 17854885
- [Background] Tetanus vaccines: WHO position paper - February 2017. Wkly Epidemiol Rec. 2017 Feb 10;92(6):53-76. No abstract available. English, French. PMID 28185446
- [Background] Yu Chao, Xu Yuming, Xu Jin, et al. Progress of clinical application and safety of tetanus antitoxin. Chinese Journal of Pharmacovigilance, 2016, 13 (1): 36-41.
- [Background] Perey BJ. Progress in tetanus prophylaxis: the advent of human antitoxin. Can Med Assoc J. 1966 Feb 26;94(9):437-41. PMID 5902706
- [Background] Plotkin, S.A., W.A. Orenstein and P.A. Offit, Plotkin's vaccines. Seventh edition. ed. 2018. 1691.
- [Background] Ortiz JR, Hombach J. Announcing the publication of the WHO immunological basis for immunization series module on influenza vaccines. Vaccine. 2018 Sep 5;36(37):5504-5505. doi: 10.1016/j.vaccine.2017.09.010. Epub 2017 Oct 16. PMID 29042200
- [Background] Forrat R, Dumas R, Seiberling M, Merz M, Lutsch C, Lang J. Evaluation of the safety and pharmacokinetic profile of a new, pasteurized, human tetanus immunoglobulin administered as sham, postexposure prophylaxis of tetanus. Antimicrob Agents Chemother. 1998 Feb;42(2):298-305. doi: 10.1128/AAC.42.2.298. PMID 9527776
- [Derived] Liang Z, Liu S, Guo W, Deng Z, Bin W, Yu A, Hu J, Wu L, Li Z, Huang W, Li H, Cheng D, Li S, Guo Q, Zhang D, Yan X, Wang C, Cai W, Ding B, Li W, Li X, Xu B, He L, Ouyang Y, Zhan H, Wang J, Zhao Y, Liu X, Xiang W, Zhang M, Zhang Z, Ding J, Kuang X, Zheng W, Liao H, Wang W, Wang C. Recombinant monoclonal antibody siltartoxatug versus plasma-derived human tetanus immunoglobulin for tetanus: a randomized, double-blind, active-controlled, phase 3 trial. Nat Med. 2025 Aug;31(8):2673-2681. doi: 10.1038/s41591-025-03791-8. Epub 2025 Jul 8. PMID 40628965